CLINICAL TRIAL: NCT03332745
Title: Mechanism of Left Ventricular Decompensation Evaluation - Aortic Stenosis
Brief Title: Mechanism of Decompensation Evaluation - Aortic Stenosis
Acronym: MODE-AS
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: E161633
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Aortic Stenosis; Myocardial Fibrosis; Left Ventricular Hypertrophy
Keywords: Troponin
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma samples Myocardial biopsy specimens Aortic valve tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe aortic stenosis: Patients with severe aortic stenosis who are scheduled to undergo aortic valve replacement surgery
- Control group: Patients scheduled to undergo non-aortic valve cardiac or elective ascending aortic surgery

SUMMARY:
Aortic stenosis is the most common heart valve disease requiring intervention in high income countries. It is characterised by progressive valvular thickening, and restriction as well is hypertrophy and fibrosis of the left ventricle in response to pressure overload. The pathological processes in the left ventricle that ultimately result in heart failure and death are incompletely understood. Further elucidation of these processes and how they correlate with novel blood biomarkers may help us design new treatments and optimise the timing of surgical intervention.

In brief, recruited patients with severe aortic stenosis and scheduled to undergo valve replacement surgery will be invited for some simple tests (blood sampling, ECG, echocardiogram). A septal myocardial biopsy will be taken at the time of surgery and the disease valve retained. These will be examined histologically and pathological changes compared with results obtained from ECG, echocardiogram and blood tests.

ELIGIBILITY:
* Inclusion Criteria (aortic stenosis group):
* Age over 18
* Severe aortic stenosis with planned aortic valve replacement

Inclusion Criteria (control group):

* Age over 18
* Planned non-aortic valve cardiac or elective ascending aorta surgery

Exclusion Criteria (aortic stenosis group):

* Coexistent severe aortic or mitral regurgitation
* Coexistent mitral stenosis greater than mild in severity
* Acute valvular heart disease (e.g. acute mitral regurgitation or endocarditis)
* Acute pulmonary oedema or cardiogenic shock
* Coexistent hypertrophic cardiomyopathy
* Unable to give informed consent

Exclusion Criteria (control group):

* Significant aortic valve disease (mild aortic stenosis / regurgitation or greater)
* Acute valvular heart disease (e.g. acute mitral regurgitation or endocarditis)
* Acute pulmonary oedema or cardiogenic shock
* Coexistent hypertrophic cardiomyopathy
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for surgery for aortic valve disease (aortic stenosis group) and those referred for non-aortic valve cardiac surgery or elective ascending aorta surgery (control group)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation of blood biomarkers with pathological changes on myocardial biopsy | Biomarkers collected within 1 month prior to date of surgery (and myocardial biopsy)
  Correlation between biomarkers (e.g. high sensitivity troponin I, BNP) with levels of myocardial fibrosis (collagen volume fraction as measured by picrosirius red staining)

SECONDARY OUTCOMES:
Correlation of echocardiographic and ECG measures with pathological changes on myocardial biopsy | Biomarkers collected within 1 month prior to date of surgery (and myocardial biopsy)
  Correlation between imaging measures (e.g. LV diastolic function, longitudinal systolic function, ECG LVH criteria, ECG strain pattern) with levels of myocardial fibrosis (collagen volume fraction as measured by picrosirius red staining)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J Everett, MBBS, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh / NHS Lothian, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided